CLINICAL TRIAL: NCT06778746
Title: Use of Biologics for Severe Asthma in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Head of Respiratory Medicine (clinical service), Chinese University of Hong Kong
Other Study IDs: CUHK_biologics_01
Record Dates: First submitted 2024-12-26; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no interventions — No interventions, this is an observational study
  Other Names: No interventions, this is an observational study

SUMMARY:
The landscape of biologics therapy used in Hong Kong is currently unknown. The purpose of this study is to conduct a retrospective analysis of the use of biologics treatment for severe asthma in Hong Kong. The study aims to assess the landscape of biologics usage, evaluate the characteristics and conditions of patients before and after receiving biologic therapy, and provide insights into the effectiveness and safety of these treatments in the local population.

DETAILED DESCRIPTION:
This is a multi-centre retrospective study of subjects using biologics for the treatment of asthma.

This study will be a retrospective, observational study utilizing data from medical records.

The investigators surveyed all subjects with asthma subjects treated by biologics used in Hong Kong from CDARS or from patient lists drawn from local pharmacies of participating hospitals. Patients' electronic and paper medical records will be reviewed by the co-investigators at the respective hospital (respiratory physicians). Name list of the patients will be drawn from 2003 when the first biologic omalizumab was approved for asthma patient use. The search period lasts till January 2024.

The identity card numbers of the patients will not be included in the database, and patients will be identified by number codes. No personal identifiable information will be reported. No patient consent would be required as this is a healthcare record study.

This study will be conducted in accordance with the principles of the Declaration of Helsinki and local ethical guidelines.

The following information will be collected:

1. The name of the biologic started
2. Indications for starting biologics
3. Date of starting (switching and stopping with dates, if any, reason for switching and stopping)
4. Demographic characteristics of the study including age, gender, body weight, body height, exposure to triggers (smoking, workplace exposure, allergens)
5. Comorbidity assessments including:

   * Old PTB
   * COPD
   * Heart Failure
   * Hypertension
   * Diabetes Mellitus
   * Hyperlipidaemia
   * Ischemic Heart Disease
   * OSA
   * Eczema
   * GERD
   * Nasal polyposis
   * Rhinitis
   * Psychiatric disorder
   * NSAID sensitivity
   * Others
6. Blood eosinophil count

   * latest one before starting biologics
   * also record the highest level in the 12 months with date preceding the commencement of biologic
   * the latest level with date
7. IgE levels

   * latest one before starting biologics
   * also record the highest level in the 12 months with date preceding the commencement of biologic
   * the latest level with date
8. Baseline spirometry (before starting biologics) and latest lung function with dates (including history of significant bronchodilator reversibility)
9. Baseline FeNO (before starting biologics) and latest FeNO with dates (also record the highest level of FeNO with date in the 12 months preceding the commencement of biologic)
10. Asthma control with estimation of ACT and GINA asthma control before and after (at 6 months, 1 year and the latest) biologic therapy with dates
11. Skin prick test results or blood allergen sensitization test results, if available
12. Age of onset of asthma
13. Number of exacerbations 12 months before starting the biologics and also exacerbations after starting the biologics (with dates at the start of the exacerbations)
14. Predominant symptom for asthma before the start of biologics
15. Medications used before and after (at 6 months, 1 year and the latest) starting biologics (including systemic corticosteroids and inhaled corticosteroids) with dates
16. Funding of the biologics (e.g. self-paid, government servants, paid by employer, paid by insurance, paid by Samaritan Fund[full/partial])
17. Any complications of steroid toxicity, including osteoporosis, fractures, obesity, DM
18. GP visits, government general outpatient visits, specialist outpatient visits, emergency department visits, hospitalizations, number of days of sick leaves taken 12 months before and after the start of biologics
19. Side effects of biologics
20. Estimation of treatment adherence (From prescription records, patients' claims, physicians' 'feel' and/or FeNO level monitoring)
21. Inhaler technique (any checking and if yes, is the technique correct)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Patients diagnosed with severe asthma per the Global Initiative for Asthma (GINA) guidelines.
* Patients who have received biologic therapy for treatment of asthma (including those who received just one dose to allow assessment of the reason for withdrawal)

Exclusion Criteria:

- Patients with respiratory diseases with other known significant respiratory diseases, including tuberculosis (TB)-destroyed lung parenchyma, history of lung resection and lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We surveyed all subjects with asthma subjects treated by biologics used in Hong Kong from CDARS or from patient lists drawn from local pharmacies of participating hospitals. Patients' electronic and paper medical records will be reviewed by the co-investigators at the respective hospital (respiratory physicians).
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
To determine the prevalence and patterns of biologics utilization for severe asthma in Hong Kong. | 12 months
  The usage of different biologics in percentages in the population of severe asthma is being studied.
To evaluate exacerbation rates before and after the initiation of biologic treatment. | 12 months
  The number of exacerbations requiring systemic steroids before and 12 months after treatment with biologics.
To evaluate the asthma control before and after the initiation of biologic treatment. | 12 months
  The asthma control was assessed using the asthma control test and GINA classification before and 12 months after treatment with biologics.
To evaluate the lung function before and after the initiation of biologic treatment. | 12 months
  The changes in FEV1 percentage predicted before and 12 months after treatment with biologics.
To explore whether physicians are following international guidelines for the prescription of biologics | baseline
  Assess the percentage of patients with biologics were prescribed according to the Global Initiative for Asthma criteria.
To identify any adverse events associated with biologic therapy in the study population | 12 months
  To assess any adverse events (including but not limited to headache, rash, allergic reaction, sore throat, tiredness) after using the biologics in 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fanny WS Ko, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, Shatin, NT, HK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No